CLINICAL TRIAL: NCT00718458
Title: EEG-Based Brain-Computer Interface Project for Individuals With ALS
Brief Title: EEG-Based Brain-Computer Interface Project for Individuals With Amyotrophic Lateral Sclerosis (ALS)
Acronym: BCI
Status: Completed | Type: Observational
Sponsor: Drexel University College of Medicine (Other)
Collaborators: MDA/ALS Center of Hope (Other)
Responsible Party: Sponsor
Organization: Drexel University (Other)
Other Study IDs: Internal-17016
Record Dates: First submitted 2008-07-14; First posted 2008-07-18 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Amyotrophic Lateral Sclerosis; Neurodegenerative Disease; Motor Neuron Disease
Keywords: Amyotrophic Lateral Sclerosis; Cerebrospinal Fluid; Neurodegenerative Disease; Motor Neuron Disease; Autonomic Nervous System; Neurodegenerative Diseases; Movement Disorders
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neurodegenerative Diseases; Motor Neuron Disease; Movement Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ALS: Subjects having either definite or probable ALS by El Escorial Criteria.
- Non-ALS: Subjects not having either definite or probable ALS by El Escorial Criteria.

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a progressive neuromuscular condition characterized by weakness, muscle wasting, fasciculations and increased reflexes. Depending on the site of onset, individuals with ALS progressively lose control of their skeletal muscles; bulbar or the extremities. As symptoms worsen and spread, muscle atrophy becomes apparent and upper motor neuron symptoms such as spasticity complicate gait (in lower limb involvement) and manual dexterity (in upper limb involvement). The patients progress to a state of profound disability and have great difficulty in communicating; some may even be entirely "locked in" to their bodies. The capacity for simple communication could greatly improve their quality of life.

New technologies are giving people with disabilities alternate communication and control options. One such instrument is the EEG-based Brain-Computer Interface (BCI) which can provide both communication and control functions to those who have lost muscle control. By recording electroencephalographic (EEG) signals or brain waves from the scalp and then decoding them, the Wadsworth BCI allows people to make selections on a computer screen [i] In this study we will be investigating the feasibility of using EEG-based Brain-Computer Interface technology as a communication solution for individuals with ALS. The specific question addressed will be: Can individuals with ALS use the BCI for communication when they present with extreme loss of neuromuscular control and severe communication impairments? The goal of the project is to determine whether this device is a practical and realistic means for individuals with ALS to communicate. The study is intended to evaluate both the complexity of the system and the degree to which each participant will be able to communicate. Trials will consist of asking the subject to follow a series of simple instructions and complete certain tasks while using the BCI.

This study design requires that the individual live in the Philadelphia region. Please contact the Wadsworth Center of the New York State Department of Health and State University of New York at Albany directly if you reside outside of this area.

DETAILED DESCRIPTION:
This study design requires that the individual live in the Philadelphia region. Please contact the Wadsworth Center of the New York State Department of Health and State University of New York at Albany directly if you reside outside of this area.

ELIGIBILITY:
Inclusion Criteria:

Medical Subjects:

* Be able to give consent themselves or via a legally authorized representative.
* Diagnosed with a neuromuscular disease and have limited ability to communicate.
* Be able to see visual cues such as targets or letters presented on the screen, and/or ability to hear auditory cues such as tones or words presented through speakers or earphones.
* Be able to understand and remember instructions concerning participation.

Healthy control subjects:

* Be able to consent to give consent themselves or via a legally authorized representative.
* Be able to see visual cues such as targets or letters presented on the screen, and/or ability to hear auditory cues such as tones or words presented through speakers or earphones.
* Be able to understand and remember instructions concerning participation.

Exclusion Criteria:

* Individuals with cognitive impairments that would impact their ability to follow the instructions

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ALS clinic patients at MDA/ALS Center of Hope.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2007-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
BCI Accuracy | 1 session
  Measurement of percent spelling accuracy of the BCI system will be a main factor in determining usability of the system.

CONTACTS AND LOCATIONS:
Overall Officials: Terry Heiman-Patterson, MD, Principal Investigator — MDA/ALS Center of Hope
Locations (1):
- MDA/ALS Center of Hope, Philadelphia, Pennsylvania, United States